CLINICAL TRIAL: NCT00439387
Title: Imaging Serotoninergic Neurotransmission in Epilepsy
Brief Title: The Role of Serotonin in Seizures
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070103; 07-N-0103
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-06-05

CONDITIONS: Epilepsy; Seizures
Keywords: Serotonin; Epilepsy; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy; Seizures

SUMMARY:
This study will investigate the role that a brain chemical called serotonin plays in seizures. Serotonin, present naturally in the brain, helps transmit signals between nerve cells. Glucose is a sugar that is the main fuel of the brain. Studying these two chemicals may help explain why people with epilepsy get seizures and are more likely to be depressed.

Healthy volunteers and patients 18 to 60 years of age who have epilepsy with or without depression and whose seizures are not controlled by medication may be eligible for this study. Candidates are screened with a review of their medical history, a physical examination and an electroencephalogram (EEG, brain wave recording).

Participants undergo the following procedures:

* Positron emission tomography (PET) scans: The first of three PET scans measures brain blood flow and the activity at some of the brain serotonin receptors (the parts of brain cells to which serotonin attaches). A second scan measures the amount of serotonin transported between brain cells. A third scan measures glucose use. The PET scanner is shaped like a doughnut. The subject lies on a bed that slides in and out of the scanner with his or her head inside the opening. A special mask is fitted to the subject s head to help keep it still during the procedure so the images will be clear. For the first scan, catheters (plastic tubes) are placed in an arm vein to inject a radioactive substance and in an artery in the wrist to collect blood samples. The other two scans require only the catheter in the arm.
* Magnetic resonance imaging: This test uses a strong magnetic field and radio waves to obtain images of the brain. The scanner is a metal cylinder surrounded by a strong magnetic field. The subject lies on a table that can slide in and out of the cylinder. Most scans last between 45 and 90 minutes. Subjects wear earplugs to muffle loud knocking noises that occur during scanning.
* Psychological evaluation: Subjects are interviewed and fill out questionnaires to help study sadness and depression in epilepsy.
* Blood draw: Blood tests look for differences in genes between people with epilepsy who are depressed and those who are not.

DETAILED DESCRIPTION:
Objective: To study serotonergic transmission in epilepsy and its relation to cerebral glucose metabolism, mesial temporal sclerosis, and depression.

Study population: Patients with localization-related epilepsy with and without depression, and generalized epilepsy, and normal controls, ages 18-60.

Design: This is a neuroimaging study using positron emission tomography with a 5HT(1A) receptor ligand, 18F-FCWAY, a serotonin transporter ligand, 11C-DASB, and 15O-H2O for cerebral blood flow estimation. Patients will have measurements of cerebral glucose metabolism using 18F-FDG as well. Magnetic resonance imaging will be performed for examination of hippocampal structure and partial volume correction. Screening for depression will be performed by NIMH investigators. We will measure cortisol and ACTH levels, which may affect hippocampal structure and function. Testing for genetic markers that may predict serotonin transporter activity and depression will be performed.

Outcome measures: 5HT(1A) receptor binding, serotonin transporter activity, cerebral blood flow, and, in patients, glucose metabolism and hippocampal structure. Patients will be stratified by seizure type and depression ratings.

ELIGIBILITY:
* INCLUSION CRITERIA:

  * Patients must have seizures documented by appropriate clinical and laboratory studies . This criterion will be established by studies performed by the referring physicians, preliminary screening in the NINDS Clinical Epilepsy Section outpatient clinic, or if necessary, inpatient video-EEG monitoring.
  * Male and Female subjects aged between 18 and 60 years
  * Healthy control subjects will also be recruited.
  * Subjects must be able to give written informed consent prior to participation in this study.

EXCLUSION CRITERIA:

* Patients younger than 18 or older than 60 years old. There is evidence for reduced 5HT1A receptor binding in patients over 60.
* Patients with a known treatable seizure etiology such as neoplastic or infectious disease.
* Patients with MRI findings consistent with brain tumors, trauma or AVMs.
* Patients with progressive neurologic disorders.
* Patients with a history of significant medical disorders, or requiring treatment with drugs

that can not be stopped, and would interfere with the study, except for antidepressants.

* Patients with cancer.
* Patients not capable of giving an informed consent.
* Patients who had seizure activity 24 hours prior to the study.
* Women who are pregnant or nursing
* Subjects who are current smokers, and cannot stop for at least two weeks before the PET scan, as smoking may affect serotonergic neurotransmission.
* Healthy subjects must be free from a personal history of seizure disorders
* Patients with coagulation abnormalities.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-02-20; Study Completion 2015-06-05

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bromfield EB, Altshuler L, Leiderman DB, Balish M, Ketter TA, Devinsky O, Post RM, Theodore WH. Cerebral metabolism and depression in patients with complex partial seizures. Arch Neurol. 1992 Jun;49(6):617-23. doi: 10.1001/archneur.1992.00530300049010. PMID 1596197
- [Background] Kanner AM. Depression in epilepsy: prevalence, clinical semiology, pathogenic mechanisms, and treatment. Biol Psychiatry. 2003 Aug 1;54(3):388-98. doi: 10.1016/s0006-3223(03)00469-4. PMID 12893113
- [Background] Lambert MV, Robertson MM. Depression in epilepsy: etiology, phenomenology, and treatment. Epilepsia. 1999;40 Suppl 10:S21-47. doi: 10.1111/j.1528-1157.1999.tb00884.x. PMID 10609603